CLINICAL TRIAL: NCT02076997
Title: Individualized High Dose Methotrexate for the Treatment of Malignancies in Children and Adolescents With a Significant Risk for Methotrexate Toxicities
Brief Title: Individualized High Dose Methotrexate to Treat Cancer in Children Who Have a Significant Risk for Side Effects to Methotrexate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Texas Children's Cancer Center (Other)
Responsible Party: Principal Investigator, Jennifer Foster, Assistant Professor of Pediatrics, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-33119
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Results first posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Cancer
Keywords: Cancer; High Dose Methotrexate
MeSH Terms: conditions — Neoplasms | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Individualized High Dose Methotrexate (Experimental): Individualized high dose methotrexate given as a 24-hour infusion.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — Patients will receive 5g/m^2 high dose methotrexate as a 24 hour infusion.
  The methotrexate level in the blood will be checked at two times during the 24-infusion. The dose will be reduced based on the level in the blood.

SUMMARY:
Pediatric cancer patients are being asked to take part in this study who have a cancer that is treated with high doses of the drug methotrexate (MTX). In addition, these patients have either had significant side effects to methotrexate in the past or their doctor thinks that they are at high risk for side effects from receiving methotrexate. Methotrexate is a cancer-fighting drug that is very important in the treatment of leukemia.

In this study, investigators are testing a new method of giving high dose methotrexate to cancer patients which may reduce the chances that the level of methotrexate in the blood is too high. When the levels are too high this is thought to lead to an increase in side effects. Side effects are unintended and unwanted results of treatment.

The initial ordered amount of methotrexate and the period over which methotrexate is given will not change from the current standard of care (meaning what is usually done by doctors, and would likely be done if the patient was not on this study). This study is testing a new method of monitoring and potentially adjusting the final amount of methotrexate that the patient will end up receiving based on levels of methotrexate in the blood in the first 24 hours in order to try to prevent side effects in patients with a previous history of side effects from methotrexate or who are at high risk for having side effects.

On this study the investigators will check methotrexate levels in the blood 2 hours after the patient starts receiving the drug and the investigators will lower the dose of methotrexate if needed. Investigators will do the same thing again 6-8 hours later.

Investigators will also collect an optional blood sample from the patient because the investigators want to study how genetic (DNA) differences are involved in how the body processes methotrexate.

DETAILED DESCRIPTION:
The study participant will receive the drug methotrexate as a patient in the hospital. High dose methotrexate will be given as a 24-hour infusion as part of the care determined to be necessary by their doctor. Infusion means the drug is given using a needle or tubing inserted into a vein (also called IV).

The standard of care in patients receiving high dose methotrexate is to give the entire dose of methotrexate, without adjustment, and to then check the concentration of methotrexate in the blood at the end of the infusion. Most patients will have a level of methotrexate in their blood which is good to treat cancer and keep side effects at a minimum. However, other patients have a level of methotrexate at the end of the 24-hour infusion which is very high and is thought to lead to an increase in side effects.

In this study, investigators are testing a method of giving methotrexate which may reduce the chances that the level of methotrexate in the blood at the end of the infusion is too high. This will be done by checking the methotrexate level in the blood at two times during the 24-hour infusion and reducing the dose of methotrexate being given if the levels are not thought to be in the correct range (the level is too high). Reducing the dose may result in the patient receiving a lower total dose of methotrexate than initially ordered. However, it may also result in a more preferred concentration of methotrexate in the blood at the end of the infusion.

It is possible that in the past the patient's doctor may have chosen to reduce the amount of methotrexate given because the patient had side effects. In this study, all patients will start out receiving the standard dose of methotrexate. Therefore, by participating in this study, the amount of methotrexate ordered at the start of the infusion may be higher than what the patient received previously.

Before and after the patient receives high dose methotrexate, the patient will receive IV fluids. In order to minimize side effects, methotrexate levels will also be closely monitored after the infusion and the patient will receive supportive medicines as needed. The patient will receive the drug Leucovorin (administered by mouth every 6 hours for minimum of 3 doses). The monitoring and supportive care that the patient will receive at the end of the methotrexate infusion, the amount of IV fluids, and the dose or duration of Leucovorin received will be done based on standard guidelines and are not part of this study.

After receiving the 24-hour high dose methotrexate, this individualized monitoring plan will end and management of the patient's methotrexate levels will continue according to standard guidelines.

High dose methotrexate may be given to the patient multiple times at the discretion of their doctor. While on this study, the patient will receive methotrexate using the methods of this study (however, they will only have blood drawn one time for optional DNA testing). The patient, his/her parent, or the doctor may decide to withdraw the patient from this study at any time if they do not think that it is in the patient's best interest to continue to receive methotrexate in the manner being investigated in this study.

STUDY RELATED TESTS AND PROCEDURES

At study entry, the following will occur:

* The patient will have a physical exam
* Collection of blood samples for routine blood tests and research blood tests. Approximately 1-2 teaspoons of blood will be taken for research blood tests.
* Review of the patient's medical and medication history to collect information.

During treatment and after treatment the following will occur:

* Collection of blood samples for routine blood tests and research blood tests. Approximately ½ teaspoon of blood will be taken at times 2, 6 (or 8), 24, 36, 42, and 48 hours. The blood collected at 2 and 6 (or 8) and 24 hours is for the research blood tests.
* Review of the patient's medical and medication history to collect information.

The research blood tests are done to see how much methotrexate is in the body, how the body handles the drug, and to do DNA studies. The DNA will be tested to look for small changes called Single Nucleotide Polymorphisms (SNP). These small changes sometimes explain why different people have different reactions to drugs. The total amount of blood drawn for the research studies is approximately 3 teaspoons.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Patients must be greater than or equal to 365 days and less than 23 years of age at the time of enrollment.
2. Diagnosis: Patients with any malignancy who will receive high dose methotrexate (HDMTX) given as a 5 g/m2 infusion over 24 hours and a history of ≥ 1 of the following:

   * Documented decreased renal function, defined as Creatinine greater than 1.5 x baseline or glomerular filtration rate (GFR) <65ml/min/1.73m2.
   * History of prior nephrotoxicity with HDMTX as evidence by increased creatinine to 1.5 x baseline or need for dialysis or carboxypeptidase
   * History of Grade 3 adverse event (AE) related to HDMTX (mucositis, myelosuppression, nephrotoxicity, hepatotoxicity) based on the NIH Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
   * Provider concern patient is at risk for MTX toxicity, such as a prior history of treatment with nephrotoxic chemotherapy, history of HDMTX-related neurotoxicity, or antimicrobial/antifungal therapy

Exclusion Criteria:

1. Unable to draw labs for HDMTX serum concentration
2. Enrollment on a protocol (COG or other) which restricts proposed dose modifications
3. Patients with Trisomy 21
4. Patients with greater than grade 1 neurologic toxicity at the time of enrollment that is attributed to unresolved prior methotrexate toxicity
5. Patients with greater than or equal to grade 3 chronic kidney disease at enrollment (eGFR or creatine clearance (CrCl) less than 30ml/min/1.73m2)

Ages: 1 Year to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2019-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer H Foster, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Derived] Foster JH, Thompson PA, Bernhardt MB, Margolin JF, Hilsenbeck SG, Jo E, Marquez-Do DA, Scheurer ME, Schafer ES. A prospective study of a simple algorithm to individually dose high-dose methotrexate for children with leukemia at risk for methotrexate toxicities. Cancer Chemother Pharmacol. 2019 Feb;83(2):349-360. doi: 10.1007/s00280-018-3733-2. Epub 2018 Nov 28. PMID 30488179

RESULTS

PARTICIPANT FLOW:
Groups:
- Individualized High Dose Methotrexate: Individualized high dose methotrexate given as a 24-hour infusion.
  Methotrexate: Patients will receive 5g/m^2 high dose methotrexate as a 24 hour infusion.
  The methotrexate level in the blood will be checked at two times during the 24-infusion. The dose will be reduced based on the level in the blood.
Period: Overall Study
Arm/Group | Individualized High Dose Methotrexate
Started | 23
Completed | 22
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Individualized High Dose Methotrexate
Number analyzed (Participants) | 22
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 13 [1 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Success (Achieving an End Infusion Peripheral Blood Methotrexate Concentration Between 50-80 μM)
Description: 1a) Calculate the incidence of success with the new protocol (achieving an end infusion peripheral blood methotrexate concentration between 50-80 μM)
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | Individualized High Dose Methotrexate
Number analyzed (Participants) | 22
uM | 57 (14)
Statistical Analysis 1: Comparison: Individualized High Dose Methotrexate; Test type: Other; p < 0.01, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Incidence of >Grade 3 Nephrotoxicity
Description: Calculate the incidence of >grade 3 nephrotoxicity
Time Frame: 2.5 months
Population: 22 patients were enrolled for a total of 54 cycles of methotrexate. Toxicities were recorded by cycle
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized High Dose Methotrexate
Number analyzed (Participants) | 54
Participants | 0

3. Secondary Outcome: Incidence of Neurotoxicity
Description: Calculate the incidence of neurotoxicity
Time Frame: 2.5 months
Population: 22 patients were enrolled for a total of 54 cycles of methotrexate. Toxicities were recorded by cycle
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized High Dose Methotrexate
Number analyzed (Participants) | 54
Participants | 1

4. Secondary Outcome: Incidence of Mucositis
Description: Calculate the incidence of mucositis
Time Frame: 2.5 months
Population: 22 patients were enrolled for a total of 54 cycles of methotrexate. Toxicities were recorded by cycle
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized High Dose Methotrexate
Number analyzed (Participants) | 54
Participants | 5

5. Secondary Outcome: Incidence of Hepatoxicity
Description: Calculate the incidence of hepatotoxicity
Time Frame: 2.5 months
Population: total infusions
Measure: Number; unit: infusions
Arm/Group | Individualized High Dose Methotrexate
Number analyzed (Participants) | 54
infusions | 10

6. Secondary Outcome: Incidence of Myelosuppression
Description: grade >/= 3 hematological toxicity
Time Frame: 2.5 months
Population: 22 patients were enrolled for a total of 54 cycles of methotrexate. Toxicities were recorded by cycle
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized High Dose Methotrexate
Number analyzed (Participants) | 54
Participants | 39

7. Other Pre Specified Outcome: Description of the Genotype of Various Methotrexate Metabolizing SNPs
Description: We described the genotype of various identified methotrexate metabolizing SNPs
Time Frame: 4 weeks
Population: The SNP analysis was descriptive data
Measure: Number; unit: percent SNPs in the population
Arm/Group | Individualized High Dose Methotrexate
Number analyzed (Participants) | 22
percent SNPs in the population
  rs1801394 | 26
  rs1801133 | 36
  rs1801131 | 29
  rs7317112 | 43
  rs4149056 | 38
Statistical Analysis 1: Comparison: Individualized High Dose Methotrexate; There was no statistical analysis performed for this aim as it was descriptive; Test type: Other; There was no statistical analysis performed for this aim as it was descriptive

8. Other Pre Specified Outcome: Examination of Predictors of Success in Achieving Goal Concentration of Methotrexate
Description: We examined the predictors of success in achieving goal concentration of methotrexate
Time Frame: 4 weeks
Population: Among subjects who required at least one dose adjustment on study (n = 14), those who carried one or two copies of the minor allele of the C677T methylenetetrahydrofolate reductase (MTHFR) gene had an OR 6.7 (95% CI 0.49-91.3) of achieving success as defined by the protocol
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Arm/Group | Individualized High Dose Methotrexate
Number analyzed (Participants) | 14
Odds Ratio | 6.7 [0.49 to 91.3]
Statistical Analysis 1: Comparison: Individualized High Dose Methotrexate; Test type: Other; Odds Ratio (OR) = 6.7

ADVERSE EVENTS:
Time Frame: Patients were followed for 4 weeks following last HDMTX or until next chemotherapy, whichever came sooner
Arm/Group | Individualized High Dose Methotrexate
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT02076997/Prot_SAP_000.pdf